CLINICAL TRIAL: NCT01068587
Title: A Phase I/II Study of Foretinib in Patients With Previously Treated Non-Small Cell Lung Cancer Receiving Standard Erlotinib Therapy
Brief Title: MET/VEGFR2 Inhibitor GSK1363089 and Erlotinib Hydrochloride or Erlotinib Hydrochloride Alone in Locally Advanced or Metastatic NSCLC That Has Not Responded to Previous Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I196; CAN-NCIC-IND196 (Other: PDQ); GSK-CAN-NCIC-IND196 (Other: GlaxoSmithKline)
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Erlotinib (Active Comparator)
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis
- Foretinib plus Erlotinib (Active Comparator)
  Interventions: Drug: MET/VEGFR2 inhibitor Foretinib; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: MET/VEGFR2 inhibitor Foretinib — PhaseI and Phase II Arm A:
  Foretinib PO daily dosing starting cycle 1 day 15 and erlotinib PO daily dosing starting cycle 1 day 1. Recommended Phase II dose to be determine in Phase I.
  Arms: Foretinib plus Erlotinib
Drug: erlotinib hydrochloride — erlotinib PO daily dosing starting cycle 1 day 1. Recommended Phase II dose to be determine in Phase I.
Other: laboratory biomarker analysis — Tumour markers alone cannot be used to assess objective tumour response. If markers are initially above the upper normal limit, however, they must normalize for a patient to be considered in complete response

SUMMARY:
RATIONALE: MET/VEGFR2 inhibitor Foretinib and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This randomized phase I/II trial is studying the side effects of erlotinib hydrochloride when given together with or without MET/VEGFR2 inhibitor Foretinib and to see how well it works in treating patients with locally advanced or metastatic non-small cell lung cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the recommended phase II dose of MET/VEGFR2 inhibitor Foretinibin combination with standard erlotinib hydrochloride therapy in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) after failure of at least one prior chemotherapy regimen, and whose EGFR-expression status is positive or unknown.
* To determine the safety, tolerability, toxicity profile, dose-limiting toxicities, and pharmacokinetic profile of MET/VEGFR2 inhibitor Foretinib and erlotinib hydrochloride in this schedule.
* To determine the correlation, if any, between the toxicity profile and pharmacokinetics.
* To assess the anti-tumor activity of MET/VEGFR2 inhibitor Foretinib in combination with erlotinib hydrochloride as evidenced by response rates, clinical benefit (complete or partial response or stable disease ≥ 8 weeks duration), and an exploratory endpoint of early assessment of tumor size as a continuous variable (when compared to erlotinib hydrochloride alone).
* To assess one-year survival rate in these patients.
* To investigate the correlation, if any, between response and biomarkers, including EGFR gene mutation, EGFR gene amplification, EGFR gene polymorphisms, c-Met gene mutation, amplification and expression, phospho-c-Met expression, K-Ras gene mutation, and baseline serum HGF levels.

OUTLINE: This is a multicenter, dose-escalation phase I study of MET/VEGFR2 inhibitor Foretinib followed by a randomized, open-label phase II study.

* Phase I (dose-escalation) : Patients receive oral erlotinib hydrochloride once daily on days 1-28. Patients receive oral MET/VEGFR2 inhibitor GSK1363089 once daily on days 15-28 during course 1 and on days 1-28 during all other courses. Courses repeat every 28 days until the maximum-tolerated dose of MET/VEGFR2 inhibitor Foretinib is determined.

Blood samples are collected on days 14 and 28 of course 1 for pharmacokinetics and day 1 of courses 1 and 2 and post treatment for pharmacodynamic studies.

* Phase II: Patients are randomized to 1 of 2 treatment arms:

  * Arm I (MET/VEGFR2 inhibitor Foretinib and erlotinib hydrochloride): Patients receive oral MET/VEGFR2 inhibitor Foretinib (at the recommended phase II dose determined in phase I) once daily and oral erlotinib hydrochloride once daily on days 1-28. Courses repeat very 28 days in the absence of disease progression or unacceptable toxicity.
  * Arm II (erlotinib hydrochloride only): Patients receive oral erlotinib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

In both arms, samples are collected for pharmacodynamic studies as in phase I.

After completion of study treatment, patients are followed at week 4 and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), meeting all of the following criteria:

  * Locally advanced or metastatic disease
  * Failed 1-2 prior chemotherapy regimen

    * Must be eligible to receive erlotinib therapy (i.e., patients must have received 1-2 prior chemotherapy regimen [combination unless patient is ≥ 70 years]) for advanced or metastatic disease
    * No plan to receive further palliative cytotoxic chemotherapy
* EGFR-expression status positive or unknown

  * Patients who are known to have tumors that are EGFR negative on IHC are not eligible
* Presence of clinically and/or radiologically documented measurable disease

  * At least 1 site of disease must be unidimensionally measurable as follows:

    * Chest X-ray ≥ 20 mm
    * CT scan (with slice thickness of ≤ 5 mm) ≥ 10 mm (longest diameter)
    * Physical exam (using calipers) ≥ 10 mm
    * Lymph nodes by CT scan ≥ 15 mm (measured in short axis)
  * Measurable lesions must be outside a previous radiotherapy field unless disease progression has been documented
* Must have archival tissue available or undergo a biopsy or FNA prior to registration/ randomization
* No appreciable cavitation in central thoracic lesions

  * Patients with overt bleeding from any site (> 30 mL bleeding/episode) within 3 months of study entry are not eligible
* No untreated brain or meningeal metastases (CT scans are not required to rule this out unless there is a clinical suspicion of CNS disease)

  * Patients with treated and radiologic or clinical evidence of stable brain metastases, with no evidence of cavitation or hemorrhage in the brain lesion, are eligible providing that they are asymptomatic and do not require corticosteroids (must have discontinued steroids ≥ 1 week prior to entry)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Patients must have discontinued smoking for ≥ 2 weeks prior to registration, and must be prepared to refrain from cigarette usage until completion of the pharmacokinetic sampling at the end of study course 1 (approximately 6 weeks in total) (Phase I only)
* Granulocyte count (AGC) ≥ 1.5 times 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Serum creatinine ≤ 1.5 times upper normal limit (UNL) OR calculated creatinine clearance ≥ 50 mL/min (≥ 0.83 mL/sec)
* Bilirubin ≤ 1.5 times UNL
* ALT and AST ≤ 2 times UNL
* No clinically relevant hemoptysis (> 5 mL fresh blood) within 4 weeks prior to study entry

  * Patients with only flecks of blood in sputum are permitted
* No other invasive malignancies, unless curatively treated with no evidence of disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 90 days after completion of study therapy
* No untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction, including any of the following:

  * Unstable angina, congestive heart failure, or myocardial infarction within the previous year
  * Cardiac ventricular arrhythmias requiring medication
  * History of 2nd or 3rd degree atrioventricular conduction defects
* Patients with a significant cardiac history (even if controlled) or prior doxorubicin exposure are required to have a LVEF > 50%
* Patients with proliferative diabetic retinopathy, retinal arteritis, or hemorrhage must undergo full ophthalmological examination prior to entry to this study
* Must have resting systolic BP ≤ 150 mm Hg and/or diastolic BP ≤ 100 mm Hg (in the presence or absence of a stable dose of anti-hypertensive medication)
* No poorly controlled hypertension
* No history of labile hypertension or poor compliance with anti-hypertensive medication
* No GI tract disease resulting in an inability to absorb oral medication, including any of the following situations:

  * Uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)
  * Post-surgical malabsorption characterized by uncontrolled diarrhea that results in weight loss and vitamin deficiency or requires IV hyperalimentation (use of pancreatic enzyme supplementation is allowed)
* No active or uncontrolled infections
* No serious illnesses or medical conditions that would not permit the patient to be managed according to the protocol
* No known hypersensitivity to the study drugs or their components

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than two prior chemotherapy regimens for metastatic NSCLC (excluding adjuvant chemotherapy)
* Recovered from any treatment-related toxicities prior to randomization

  * Persistent cisplatin- or taxane-induced sensory neuropathy ≤ grade 2 is acceptable
* No prior therapy with agents acting on the EGFR pathway
* No prior therapy with a c-Met inhibitor
* At least 21 days since the last dose of chemotherapy
* At least 21 days since last fraction of prior radiation therapy

  * Exceptions may be made for non-myelosuppressive radiation to peripheral areas
* More than 14 days since prior major surgery, provided that wound healing has occurred
* More than 3 weeks since prior and no other concurrent investigational drugs or anti-cancer therapy
* No concurrent CYP3A4 enzyme inducing or inhibiting drugs known to interact with erlotinib hydrochloride, including any of the following:

  * Enzyme-inducing anticonvulsants
  * Rifampicin
  * Rifabutin
  * St. John wort
  * Atazanavir
  * Ketoconazole
* Patients with a history of pulmonary embolus or a deep vein thrombosis diagnosed and/or treated within 6 months prior to registration will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-01-21 (Actual); Primary Completion 2014-03-21 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
The recommended phase II dose of daily oral MET/VEGFR2 inhibitor Foretinib when given in combination with standard erlotinib hydrochloride therapy (phase I) | 3 years
  After completion of Phase I portion of the study
Safety, tolerability, dose-limiting toxicities, and pharmacokinetic profile (phase I) | 3 years
  Assessed from the time of first dose. Results will be analyzed at time of final analysis
Correlation between toxicity and pharmacokinetics (phase I) | 3 years
  After completion of phase I
Objective tumor response rate (partial or complete response) (phase II) | After every second cycle

SECONDARY OUTCOMES:
Clinical benefit (complete response, partial response, and stable disease for ≥ 8 weeks) (phase II) | 8 weeks
  End of every second cycle
Tumor size at 8 weeks (phase II) | 8 weeks
  At end of second cycle.
1-year survival rate (phase II) | 1 year
Response or stable disease duration (phase II) | After progression
Progression-free survival (phase II) | 3 years
  After completion of therapy
Toxicity (phase II) | 3 years
  From the time of 1st dose and will be assessed overall at the time of final analysis

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada; Cheryl Ho, MD, Study Chair — British Columbia Cancer Agency
Locations (4):
- Canada (4):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leighl NB, Tsao MS, Liu G, Tu D, Ho C, Shepherd FA, Murray N, Goffin JR, Nicholas G, Sakashita S, Chen Z, Kim L, Powers J, Seymour L, Goss G, Bradbury PA. A phase I study of foretinib plus erlotinib in patients with previously treated advanced non-small cell lung cancer: Canadian cancer trials group IND.196. Oncotarget. 2017 Jun 28;8(41):69651-69662. doi: 10.18632/oncotarget.18753. eCollection 2017 Sep 19. PMID 29050231